CLINICAL TRIAL: NCT05162651
Title: Effect of Extended Cannabis Abstinence on PTSD Symptoms
Acronym: CANPOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Ahmed N Hassan, Doctor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 087-2021
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: PTSD; Cannabis Use; Cognitive Symptom; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Neurobehavioral Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency management group (Active Comparator): Randomized to receive individual motivational interviewing therapy and contingency management
  Interventions: Behavioral: Contingency-management; Other: Enhanced usual care
- Control group (Other): Randomized to receive individual motivational interviewing therapy alone
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: Contingency-management — In addition to structured assessments at baseline, four, eight and twelve months, subjects randomized to the contingency-management group will receive a contingent bonus if the participants show successful abstinence at the end of weeks 4, 8 and 12.
  Arms: Contingency management group
Other: Enhanced usual care — Subjects will receive structured, quantitative assessments at baseline, four, eight and twelve weeks.

SUMMARY:
This will be a 12-week randomized trial. Outpatients and patients from the Mood and Anxiety program at the Centre for Addiction and Mental Health (CAMH) with a current diagnosis of post-traumatic stressed disorder (PTSD) and cannabis-use disorder (CUD) will be randomized to receive individual motivational interviewing therapy and contingency management (n = 12) or individual motivational interviewing therapy alone (control group, n = 12) after enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 55 years (from both sexes [or genders]);
2. Diagnosed with CUD (moderate or severe) according to the Structured Clinical Interview for DSM-IV (SCID) (mode of cannabis consumption can be inhalation or ingestion);
3. Diagnosis of current (past 30 days) PTSD, using the CAPS-5 on screening;
4. On antidepressant medication(s) for at least 1 month (to ensure safety and homogeneity as PTSD treatment of our population);
5. Be able to provide written informed consent; and
6. Be able to communicate in English.

Exclusion Criteria:

1. diagnosed with a severe or unstable medical illness that precludes safe participation in the study as per the study physician;
2. diagnosed with schizophrenia, schizoaffective disorder, or bipolar disorder or current acute psychosis or mania based on DSM-5 criteria;
3. current suicidality risk as indicated by the Columbia Suicide Severity Rating Scale (C-SSRS) with concurrence after the study physician's evaluation if the response to C-SSRS questions 1 or 2 is "yes" 34; and
4. have pain interfering with normal function as reported by the 12-Item Short Form Survey (SF-12) (moderate or higher interference).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Severity of PTSD symptoms, as measured with the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) at week 4 | Week 0-4
  Changes in CAPS-5 during the study phase between the group that achieved abstinence and the group that did not. In addition, we will record changes in each PTSD symptom category, which will all be part of the larger trial analysis.

SECONDARY OUTCOMES:
Changes in cognitive function, as measured with various Cambridge Automated Neuropsychological Test Automated Battery (CANTAB) cognitive tests | Week 0-4
  Changes between abstainers and non-abstainers on cognitive testing during the study phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided